CLINICAL TRIAL: NCT03817723
Title: Radiation Exposure of Intraoperative Cholangiography During Cholecystectomy
Brief Title: Radiation Exposure in Intraoperative Cholangiography
Status: Completed | Type: Observational
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Olli Helminen, M.D, Ph.D., Jyväskylä Central Hospital
Other Study IDs: Rad1
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Radiation Exposure
Keywords: Radiation dose; cholangiography; Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Specialist surgeon: Radiation exposure of intraoperative cholangiography during cholecystectomy. C-arm cholangiography is performed routinely. KAP (Kerma area product) is the product of air Kerma in the center of the imaging area multiplied with size of the imaging area. For simplicity we have unified varying units received from different c-arms and will only use Gray multiplied by square centimeters (Gycm2 ). KAP values were measured using inbuilt ionization chambers in c-arms. For this study we collected the KAP values from exposure and pulsed fluoroscopy. We also recorded the fluoroscopy time (s).
  Interventions: Radiation: c-arm cholangiography
- Resident surgeon: Radiation exposure of intraoperative cholangiography during cholecystectomy.C-arm cholangiography is performed routinely. KAP (Kerma area product) is the product of air Kerma in the center of the imaging area multiplied with size of the imaging area. For simplicity we have unified varying units received from different c-arms and will only use Gray multiplied by square centimeters (Gycm2 ). KAP values were measured using inbuilt ionization chambers in c-arms. For this study we collected the KAP values from exposure and pulsed fluoroscopy. We also recorded the fluoroscopy time (s).
  Interventions: Radiation: c-arm cholangiography

INTERVENTIONS:
Radiation: c-arm cholangiography

SUMMARY:
Aims: to determine the radiation exposure of routine intraoperative cholangiography (IOC )during cholecystectomy and examine the factors affecting radiation dose and fluoroscopy time (FT).

Methods: 598 intraoperative cholangiography examinations were performed at the Central Finland Central Hospital. In this study we included 324 intraoperative cholangiographies performed with c-arm equipment not exceeding 10 years of age.

DETAILED DESCRIPTION:
From January 2016 to December 2017, consecutive 598 intraoperative cholangiography examinations were performed at the Central Finland Central Hospital. In this study we included 353 cholangiographies, that were performed with our c-arm equipment not exceeding 10 years of age in the beginning of 2016. The main measures of outcome were the recorded radiation dose data of c-arm systems from our manual database .

Another 25 cases were excluded because it was not possible to cross-check the manually recorded radiation dose data from the Picture Archiving and Communication System (PACS ). Additional 4 patients who underwent intraoperative endoscopic retrograde cholangiopancreatography (ERCP) were removed from the radiation exposure analysis because IOC and ERCP were performed consequently with the same c-arm and the radiation exposure of IOC could not be separated from the registered total KAP and FT. Thus the final analysis consisted of 324 IOCs. KAP (Kerma area product) is the product of air Kerma in the center of the imaging area multiplied with size of the imaging area. For simplicity we have unified varying units received from different c-arms and will only use Gray multiplied by square centimeters (Gycm2 ). KAP values were measured using inbuilt ionization chambers in c-arms. For this study we collected the KAP values from exposure and pulsed fluoroscopy. We also recorded the fluoroscopy time (s).

Laparoscopic cholecystectomies were performed both by residents and specialist surgeons.

Ethics: No ethical approval or written informed consent were needed because the study was retrospective in nature. The study was approved by the hospital administration.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive intraoperative cholangiographies performed with c-arm equipment not exceeding 10 years of age between January 2016 to December 2017

Exclusion Criteria:

* intraoperative cholangiographies performed with c-arm equipment exceeding over 10 years of age between January 2016 to December 2017
* patients who underwent intraoperative endoscopic retrograde cholangiopancreatography (ERCP)
* if the manually recorded radiation dose data could not be cross-checked from the Picture Archiving and Communication System ( PACS ) system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent laparoscopic , open or conversion cholecystectomy with intraoperative cholangiography
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
mean kerma area product (KAP) | 2 years
  KAP values were measured using inbuilt ionization chambers in c-arms.

SECONDARY OUTCOMES:
mean fluoroscopy time (FT ) | 2 years
  recorded from c -arms

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mattila, M.D., Ph.D., Principal Investigator — consultant surgeon
Locations (1):
- Central Finland Central Hospital, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford JA, Soop M, Du J, Loveday BP, Rodgers M. Systematic review of intraoperative cholangiography in cholecystectomy. Br J Surg. 2012 Feb;99(2):160-7. doi: 10.1002/bjs.7809. Epub 2011 Dec 19. PMID 22183717
- [Background] Murison MS, Gartell PC, McGinn FP. Does selective peroperative cholangiography result in missed common bile duct stones? J R Coll Surg Edinb. 1993 Aug;38(4):220-4. PMID 7693932
- [Background] Tusek D, Hufschmidt M, Raguse T. [Value of intraoperative laparoscopic cholangiography]. Zentralbl Chir. 1997;122(3):153-6. German. PMID 9206908
- [Background] Hauer-Jensen M, Karesen R, Nygaard K, Solheim K, Amlie EJ, Havig O, Rosseland AR. Prospective randomized study of routine intraoperative cholangiography during open cholecystectomy: long-term follow-up and multivariate analysis of predictors of choledocholithiasis. Surgery. 1993 Mar;113(3):318-23. PMID 8441966
- [Background] Nies C, Bauknecht F, Groth C, Clerici T, Bartsch D, Lange J, Rothmund M. [Intraoperative cholangiography as a routine method? A prospective, controlled, randomized study]. Chirurg. 1997 Sep;68(9):892-7. doi: 10.1007/s001040050290. German. PMID 9410677
- [Background] Amott D, Webb A, Tulloh B. Prospective comparison of routine and selective operative cholangiography. ANZ J Surg. 2005 Jun;75(6):378-82. doi: 10.1111/j.1445-2197.2005.03393.x. PMID 15943720
- [Background] Khan OA, Balaji S, Branagan G, Bennett DH, Davies N. Randomized clinical trial of routine on-table cholangiography during laparoscopic cholecystectomy. Br J Surg. 2011 Mar;98(3):362-7. doi: 10.1002/bjs.7356. Epub 2010 Nov 24. PMID 21254008
- [Background] Rehani MM, Ciraj-Bjelac O, Vano E, Miller DL, Walsh S, Giordano BD, Persliden J. ICRP Publication 117. Radiological protection in fluoroscopically guided procedures performed outside the imaging department. Ann ICRP. 2010 Dec;40(6):1-102. doi: 10.1016/j.icrp.2012.03.001. PMID 22732420
- [Background] Greffier J, Etard C, Mares O, Pereira F, Defez D, Duverger C, Branchereau P, Beregi JP, Coulomb R, Larbi A. Patient dose reference levels in surgery: a multicenter study. Eur Radiol. 2019 Feb;29(2):674-681. doi: 10.1007/s00330-018-5600-2. Epub 2018 Aug 1. PMID 30069810
- [Background] Karthikesalingam A, Markar SR, Weerakkody R, Walsh SR, Carroll N, Praseedom RK. Radiation exposure during laparoscopic cholecystectomy with routine intraoperative cholangiography. Surg Endosc. 2009 Aug;23(8):1845-8. doi: 10.1007/s00464-008-0279-0. Epub 2009 Jan 1. PMID 19118424
- [Background] Overby DW, Apelgren KN, Richardson W, Fanelli R; Society of American Gastrointestinal and Endoscopic Surgeons. SAGES guidelines for the clinical application of laparoscopic biliary tract surgery. Surg Endosc. 2010 Oct;24(10):2368-86. doi: 10.1007/s00464-010-1268-7. Epub 2010 Aug 13. No abstract available. PMID 20706739
- [Background] Singh AN, Kilambi R. Single-stage laparoscopic common bile duct exploration and cholecystectomy versus two-stage endoscopic stone extraction followed by laparoscopic cholecystectomy for patients with gallbladder stones with common bile duct stones: systematic review and meta-analysis of randomized trials with trial sequential analysis. Surg Endosc. 2018 Sep;32(9):3763-3776. doi: 10.1007/s00464-018-6170-8. Epub 2018 Mar 30. PMID 29603004
- [Background] Moller M, Gustafsson U, Rasmussen F, Persson G, Thorell A. Natural course vs interventions to clear common bile duct stones: data from the Swedish Registry for Gallstone Surgery and Endoscopic Retrograde Cholangiopancreatography (GallRiks). JAMA Surg. 2014 Oct;149(10):1008-13. doi: 10.1001/jamasurg.2014.249. PMID 25133326
- [Background] Videhult P, Sandblom G, Rasmussen IC. How reliable is intraoperative cholangiography as a method for detecting common bile duct stones? : A prospective population-based study on 1171 patients. Surg Endosc. 2009 Feb;23(2):304-12. doi: 10.1007/s00464-008-9883-2. Epub 2008 Apr 9. PMID 18398646
- [Background] Vlek SL, van Dam DA, Rubinstein SM, de Lange-de Klerk ESM, Schoonmade LJ, Tuynman JB, Meijerink WJHJ, Ankersmit M. Biliary tract visualization using near-infrared imaging with indocyanine green during laparoscopic cholecystectomy: results of a systematic review. Surg Endosc. 2017 Jul;31(7):2731-2742. doi: 10.1007/s00464-016-5318-7. Epub 2016 Nov 14. PMID 27844236
- [Background] Jolley J, Lomelin D, Simorov A, Tadaki C, Oleynikov D. Resident involvement in laparoscopic procedures does not worsen clinical outcomes but may increase operative times and length of hospital stay. Surg Endosc. 2016 Sep;30(9):3783-91. doi: 10.1007/s00464-015-4674-z. Epub 2015 Nov 19. PMID 26585194
- [Result] Buddingh KT, Weersma RK, Savenije RA, van Dam GM, Nieuwenhuijs VB. Lower rate of major bile duct injury and increased intraoperative management of common bile duct stones after implementation of routine intraoperative cholangiography. J Am Coll Surg. 2011 Aug;213(2):267-74. doi: 10.1016/j.jamcollsurg.2011.03.004. Epub 2011 Apr 3. PMID 21459631

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03817723/SAP_000.pdf